CLINICAL TRIAL: NCT00271102
Title: Randomized Trial Comparing Anterior Colporrhaphy to Paravaginal Defect Repair for Anterior Vaginal Wall Prolapse
Brief Title: Surgical Study Comparing 2 Procedures for the Treatment of a Dropped Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-0193
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Prolapse
Keywords: Cystocele, prolapse, anterior repair, colporrhaphy
MeSH Terms: conditions — Prolapse; Cystocele

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior colporrhaphy (Active Comparator): Anterior vaginal wall colporrhaphy (repair) for cystocele (dropped bladder)
  Interventions: Procedure: anterior vaginal repair (colporrhaphy); Procedure: abdominal paravaginal defect repair
- Paravaginal defect repair (Active Comparator): Abdominal paravaginal defect repair cystocele (dropped bladder)
  Interventions: Procedure: anterior vaginal repair (colporrhaphy); Procedure: abdominal paravaginal defect repair

INTERVENTIONS:
Procedure: anterior vaginal repair (colporrhaphy) — vaginal repair
Procedure: abdominal paravaginal defect repair — abdominal repair

SUMMARY:
The purpose of this study is to determine whether vaginal repair or abdominal repair is the procedure of choice for the surgical management of a prolapsed bladder.

DETAILED DESCRIPTION:
It is not known whether anterior vaginal repair (colporrhaphy) or abdominal paravaginal defect repair is the procedure of choice for the treatment anterior vaginal wall prolapse. This randomized prospective study will attempt to answer this question by assessing the change in the stage of prolapse before and after surgery, patient satisfaction through quality of life and sexual function questionnaires before and after surgery, and peri-operative complication rates. Patients enrolled into the study will be followed up for up to 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 seen at the urogynecology clinic at Geisinger with primary or recurrent pelvic organ prolapse including an anterior vaginal wall relaxation with or without urinary incontinence who are scheduled to have pelvic reconstructive surgery will be eligible to participate in the trial.

Exclusion Criteria:

* Patients with at least 2 previous prolapse surgeries
* Patients who are pregnant or planning to have a pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-01; Primary Completion 2010-02 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vatche A Minassian, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

REFERENCES:
- [Derived] Minassian VA, Parekh M, Poplawsky D, Gorman J, Litzy L. Randomized controlled trial comparing two procedures for anterior vaginal wall prolapse. Neurourol Urodyn. 2014 Jan;33(1):72-7. doi: 10.1002/nau.22396. Epub 2013 Mar 18. PMID 23508540
- See also: Click here for more information about Clinical Trials at Geisinger Medical Center — http://www.geisinger.org/research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment were between 2006 and 2010. Patients were recruited from the urogynecology outpatient clinic at Geisinger.
Pre-assignment Details: 90 patients were screened for eligibility and 70 were recruited. The remaining 20 either declined participation or were not eligible.
Period: Overall Study
Arm/Group | Anterior Colporrhaphy | Paravaginal Defect Repair
Started | 35 | 35
Completed | 30 | 30
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anterior Colporrhaphy | Paravaginal Defect Repair | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11) | 53 (13) | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in the Stage of Prolapse of the Anterior Vaginal Wall Before and One Year After Surgery
Description: POP-Q (pelvic organ prolapse quantification) as measured after surgery at one year or more after surgery. If one year data not available, then the last post-op measure is reported.
Time Frame: 4 years
Population: Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for pre-specified Primary and Secondary Outcome Measures to report in Outcome Measure data table(s).
Groups:
- POP Q Stage: Prolapse stage at followed as measured by the POP-Q system
Arm/Group | POP Q Stage
Number analyzed (Participants) | 0

2. Secondary Outcome: The Difference in Intra-operative and Post-operative Complications. Patient Satisfaction Before and One Year After Surgery Based on Quality of Life and Sexual Function Questionnaires Specifically Designed for Patients With Pelvic Organ Prolapse.
Time Frame: 4 years
Population: as for outcome 1
Groups:
- Complications: INtra-op and post-op complications
Arm/Group | Complications
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for the time frame.
Description: Per our current document retention policy, and the fact that the investigator, study staff, and record owner are no longer employed at our site, we do not have any collected data for adverse events.
Arm/Group | Anterior Colporrhaphy | Paravaginal Defect Repair
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No